CLINICAL TRIAL: NCT01028144
Title: Self-Determination for Increasing Physical Activity
Brief Title: The Active by Choice Today (ACT) Trial to Increase Physical Activity
Acronym: ACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dawn Wilson, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00005526; R01HD045693 (NIH)
Record Dates: First submitted 2009-12-01; First posted 2009-12-09 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2009-12

CONDITIONS: Exercise; Physical Activity; Obesity
Keywords: Exercise; Physical Activity; Adolescent; Minority Health
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT Program (Experimental): Motivational and Behavioral Skills Physical activity after-school program
  Interventions: Behavioral: Physical Activity Program
- General Health (Active Comparator): General health education after-school program
  Interventions: Behavioral: General Health Program

INTERVENTIONS:
Behavioral: Physical Activity Program — A 17-week motivational and behavioral skills after-school intervention for increasing moderate to vigorous physical activity in low income and minority adolescents.
  Other Names: ACT
  Arms: ACT Program
Behavioral: General Health Program — A 17-week general health afterschool intervention (comparison program) focused on nutrition, stress management, drug prevention, and drop-out prevention.
  Other Names: Comparison
  Arms: General Health

SUMMARY:
The increasing prevalence of obesity in U.S. children and adolescents is a major health threat to our society, especially among minority and low social economic status (SES) populations. During adolescence physical activity (PA) decreases and is likely an important contributor to the increasing trend in childhood obesity rates. Little evidence suggests that school-based curriculum interventions lead to increases in overall PA. Thus, this proposal will evaluate the efficacy of an innovative motivational and behavioral skills after-school program for promoting increases PA among underserved adolescents (e.g., minorities, low SES). The motivational plus behavioral skills intervention is consistent with Self-Determination (Motivation) Theory and Social Cognitive Theory in that it emphasizes increasing intrinsic motivation and behavioral skills for PA. Adolescents in the intervention take part in developing the program, selecting physical activities that generate fun and interest, and generating their own coping strategies for making effective PA changes during a videotaped session. Preliminary data from our group demonstrates the feasibility of the motivational plus behavioral skills PA program for increasing moderate-to-vigorous PA (MVPA) in underserved adolescents in South Carolina. The proposed project will use a school-based nested cohort design to evaluate efficacy of a 17-week motivational plus behavioral skills program versus typical after-school program (general health education only) on increasing PA in underserved adolescents. Twenty-four middle schools (70 6th graders per school; N=1,680), located in South Carolina will be randomly assigned to one of two after-school programs. The study employs a nested cohort design, with schools, rather than individuals assigned to condition and will be analyzed using repeated measures analysis of covariance techniques as outlined by Murray. We will also examine psychosocial variables (PA self-efficacy, self-concept, motivation, social support, and enjoyment) as potential mediators of the intervention on changes in MVPA using regression and structural equation modeling techniques. This study will address an important public health problem that will have implications for decreasing obesity in underserved adolescents.

ELIGIBILITY:
Inclusion Criteria:

* parental consent
* agree to random assignment
* 6th grade student

Exclusion Criteria:

* medical condition that interfered with physical activity
* developmentally delayed such that the intervention materials were not cognitively appropriate
* currently in treatment for a psychiatric disorder

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1422 (Actual)
Dates: Start 2004-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
moderate to vigorous physical activity (based on accelerometry estimates) | 2 weeks post intervention

SECONDARY OUTCOMES:
moderate to vigorous physical activity during the intervention (based on accelerometry estimates) | week 8 of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Wilson, PhD, Principal Investigator — University of South Carolina; Heather E Kitzman-Ulrich, PhD, Study Director — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Background] Wilson DK, Kitzman-Ulrich H, Williams JE, Saunders R, Griffin S, Pate R, Van Horn ML, Evans A, Hutto B, Addy CL, Mixon G, Sisson SB. An overview of "The Active by Choice Today" (ACT) trial for increasing physical activity. Contemp Clin Trials. 2008 Jan;29(1):21-31. doi: 10.1016/j.cct.2007.07.001. Epub 2007 Jul 17. PMID 17716952